CLINICAL TRIAL: NCT02977546
Title: Noninvasive Pulse Contour Analysis for Hemodynamic Assessment in Patients With Chronic Heart Failure
Status: Completed | Type: Observational
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Responsible Party: Principal Investigator, Thomas Bitter, Principal Investigator, Consultant for Cardiology and Pneumology, Doctor of medicine, Heart and Diabetes Center North-Rhine Westfalia
Other Study IDs: HDZNRW-KA_008_TB
Record Dates: First submitted 2016-11-16; First posted 2016-11-30 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Heart Failure
Keywords: Hemodynamics; Noninvasive; Pulse contour analysis; Heart failure; Swan Ganz Catheterization; Pulmonary artery Catheter
MeSH Terms: conditions — Heart Failure | interventions — Catheterization, Swan-Ganz

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart Failure: Patients with chronic heart failure NYHA >= 2 based on a reduced left ventricular ejection fraction (LV-EF <= 45%). All patients receive pulmonary artery catheterization and noninvasive pulse contour Analysis.
  Interventions: Device: Noninvasive pulse contour analysis; Device: Pulmonary artery catheterization

INTERVENTIONS:
Device: Noninvasive pulse contour analysis — For noninvasive pulse contour Analysis we use the CNAP-Monitor (CNSystems Medizintechnik AG, Graz, Austria)
Device: Pulmonary artery catheterization — As a reference method we use the Goldstandard intermittent thermodilution via a PAC which is regularly performed during the patients Hospital stay

SUMMARY:
Determination of hemodynamics plays an important role in the diagnosis of chronic heart failure. The gold standard is intermittent thermodilution via pulmonary artery catheter (PAC). Because of its invasiveness, there are certain risks of this method, e.g. injuries to the nerves and vessels, excessive bleedings, pneumothorax, cardiac arrhythmias etc. Noninvasive pulse contour Analysis (NPCA) is a new method which is able to determine hemodynamics noninvasively via a simple finger cuff. Advantages towards pulmonary artery Catheterization include a lower risk and an operator-Independent easy handling. Some studies investigated the accuracy, precision and trending abilities of noninvasive pulse contour analysis during anesthesia and in the intensive care unit, but there is no data available for its use in patients with chronic heart failure. The investigators therefore initiated this Trial to verify if NPCA is suitable for Determination of hemodynamics in patients with chronic heart failure.

DETAILED DESCRIPTION:
Determination of hemodynamics plays an important role in the diagnosis of chronic heart failure. The gold standard is intermittent thermodilution via pulmonary artery catheter (PAC). Because of its invasiveness, there are certain risks of this method, e.g. injuries to the nerves and vessels, excessive bleedings, pneumothorax, cardiac arrhythmias etc. Noninvasive pulse contour Analysis (NPCA) is a new method which is able to determine hemodynamics noninvasively via a finger cuff. Advantages towards pulmonary artery Catheterization include a lower risk and an operator-Independent easy handling. Some studies investigated the accuracy, precision and trend abilities of noninvasive pulse contour analysis during anesthesia and in the intensive care unit, but there is no data for its use in patients with chronic heart failure. The investigators therefore initiated this Trial to verify if NPCA is suitable for Determination of hemodynamics in patients with chronic heart failure. For NPCA the investigators use the CNAP monitor (CNSystems Medizintechnik AG). As a reference method the investigators use intermittent thermodilution via PAC (TD). Three averaged autocalibrated NPCA-CO-measurements are going to be validated against three averaged TD-CO-measurements. Moreover, measurements of cardiac index, stroke volume, systemic vascular resistance and a between-calibration-drift will be performed. The investigators will assess the accuracy and precision of the individual values.

ELIGIBILITY:
Inclusion Criteria:

* chronic heart failure NYHA >= 2 based on a reduced left ventricular ejection fraction (LV-EF <= 45%)
* written consent

Exclusion Criteria:

* high-grade tricuspid insufficiency
* implantation of a ventricular assist device (VAD)
* NIBP difference >= 20 mmHg between left and right arm before investigation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic heart failure NYHA >= 2 based on a reduced left ventricular ejection fraction (LV-EF <= 45%).
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2016-11; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Cardiac Output (l/min) | 1 day
  Three repeated and averaged measurements in a row of both methods within a range of <= 10%

SECONDARY OUTCOMES:
Cardiac index (l/min/m2) | 1 day
  Three repeated and averaged measurements in a row of both methods within a range of <= 10%
Stroke volume (ml) | 1 day
  Three repeated and averaged measurements in a row of both methods within a range of <= 10%
Systemic vascular resistance (dyn*sec/cm5) | 1 day
  Three repeated and averaged measurements in a row of both methods within a range of <= 10%

OTHER OUTCOMES:
Between-Calibration-Drift | 1 day
  One measurement before and after a new calibration including finger change

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bitter, Dr. med., Principal Investigator — Heart and Diabetes Center NRW
Locations (1):
- Clinic for Cardiology, Herz- und Diabetszentrum NRW, Ruhr-Universität Bochum, Bad Oeynhausen, Germany

IPD SHARING:
Plan to Share IPD: No